CLINICAL TRIAL: NCT01887067
Title: Renal Denervation Therapy for Resistant Hypertension in Type 2 Diabetes Mellitus
Acronym: HTN2DM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment and change in clinical evidence
Sponsor: Pamela Youde Nethersole Eastern Hospital (Other)
Responsible Party: Principal Investigator, Kin Lam TSUI, Consultant Physician, Pamela Youde Nethersole Eastern Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HKEC-2012-038
Record Dates: First submitted 2013-06-24; First posted 2013-06-26 (Estimated); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Hypertension, Resistant; Diabetes Mellitus; Renal Denervation Therapy
Keywords: Hypertension; Diabetes Mellitus
MeSH Terms: conditions — Hypertension; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Renal denervation therapy (Experimental)
  Interventions: Procedure: Renal denervation therapy

INTERVENTIONS:
Procedure: Renal denervation therapy
  Other Names: Renal denervation using Symplicity® Catheter System™

SUMMARY:
To demonstrate the efficacy of renal denervation therapy in treating resistant hypertension and its effect on glucose metabolism in patients with type 2 diabetes mellitus

ELIGIBILITY:
Inclusion Criteria:

* Age ranges from 18 to 70 years inclusive
* Essential hypertension
* Office Systolic BP (SBP) ≥ 150 mmHg or Diastolic BP (DBP) ≥ 90mmHg
* 3 or more anti-hypertensive medications of different classes, including a diuretic, or documented intolerance to multiple medications
* Type 2 Diabetes Mellitus on oral hypoglycaemic agent (OHA)
* 2 functional kidneys; eGFR ≥ 45 mL/min/1.73m² (MDRD formula)
* Suitable renal anatomy compatible with the endovascular denervation procedure

Exclusion Criteria:

* Individual has renal artery anatomy that is ineligible for treatment including:
* Patients with secondary hypertension
* Myocardial infarction, unstable angina pectoris, cerebrovascular accident within 6 months
* Patient with type 1 diabetes mellitus
* Patient on insulin due to oral drug failure
* Renovascular abnormalities (including severe renal artery stenosis, previous renal stenting or angioplasty, or known dual renal arteries)
* Pregnancy
* Patient with any implantable device incompatible with radiofrequency energy delivery
* Hemodynamically significant valvular heart disease for which reduction of BP would be considered hazardous
* Any serious medical condition, which in the opinion of the investigator, may limit the life expectancy of patients or adversely

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-06; Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Change in office systolic & diastolic blood pressure from baseline to 6 months | 6 months

SECONDARY OUTCOMES:
Change in office systolic and diastolic blood pressure up to 3 years | 3 years
Change in insulin sensitivity | 12 months
  HOMA-IR index at baseline, 3-month and 12-month
Change in glucose metabolism | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Kin Lam Tsui, FRCP (Edin, Glasg), Principal Investigator — Pamela Youde Nethersole Eastern Hospital
Locations (1):
- Pamela Youde Nethersole Eastern Hospital, Hong Kong, Hong Kong